CLINICAL TRIAL: NCT01770782
Title: Orthodontic Retention on Dental and Skeletal Maxillary Transverse Stability After Surgically Assisted Rapid Maxillary Expansion (SARME)Using Laser Scanner
Brief Title: Orthodontic Retention on the Maxillary Stability After SARME Using Laser Scanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Domingues Pereira (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Max Domingues Pereira, MD, PhD, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0949/09
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2009-07

CONDITIONS: Maxillary Hypoplasia
Keywords: Palatal Expansion Technique; Orthognathic Surgery; Three Dimensional images
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser Scanner (Other): Laser Scanner (Vivid 9i® - Konica Minolta)was used to digitize the study casts. After scanning the dental casts a 3D virtual dental casts was used to realize all measurements (pre-treatment, 4 months and 10 months).
  Interventions: Other: Laser Scanner
- SARME (Other): Surgically Assisted rapid Maxillary Expansion -SARME was used for the treatment of transverse maxillary deficiency.This procedure is a combination of a surgical procedure and orthopedic expansion of the maxilla.
  Interventions: Procedure: Surgically Assisted Rapid Maxillary Expansion (SARME)

INTERVENTIONS:
Procedure: Surgically Assisted Rapid Maxillary Expansion (SARME) — Surgical technique is performed with subtotal LeFort I osteotomy with separation of the pterygomaxillary fissure.The procedure was performed under general anesthesia using endotracheal intubation. Following the osteotomies, the expander screw was activated to 1.6 mm intraoperatively until a small diastema was observed between the upper central incisors. The incision was sutured along two planes.
  Arms: SARME
Other: Laser Scanner — Laser Scanner Vivid 9i was used to digitize the study models. The 3d virtual dental casts is a reliable copy of the original dental casts. On this virtual casts all measurements (linear, area and volume of the palate) was done to evaluate the stability after SARME.
  Arms: Laser Scanner

SUMMARY:
The objective of this study was to evaluate the effect of the orthodontic retainer on transverse maxillary dental and skeletal stability after SARME.

DETAILED DESCRIPTION:
Methods: Ninety digitized dental casts of 30 adult patients (18 males and 12 females) submitted to SARME using the Hyrax expansion appliance were evaluated. Patients were distributed into two groups: Group Without Retention (GSC) n = 15; and Group With Retention (GCC) n = 15. In the GCC group, a Transpalatal Arch (TPA) was installed for retention soon after removal of the expander. The dental casts were scanned using a Vivid 9i 3D laser scanner (Konica Minolta, Wayne, NJ). The plaster models were performed preoperatively (T1), 4 months after the expander was removed (T2), and 10 months after the end of the expansion (T3). The distances measured were Inter-Cusps of Premolars and Molars (Inter-Cusp PM) (Inter-Cusp M), Inter-Cervicals of Premolars and Molars (Inter-Cervical PM) (Inter-Cervical M), Inter-WALA edges of Premolars and Molars (PM Inter-BW) (BW Inter-M), palatal height at the molar, and palatal area and volume at T1, T2, and T3.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with bilateral transverse maxillary deficiencies greater than 5 mm

Exclusion Criteria:

* Patients with previous histories of maxillary surgery,
* congenital craniofacial malformations and
* unilateral transverse maxillary deficiencies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maxillary Stability | up to 10 months after the end of expansion
  Laser scanner to create a 3D virtual dental cast

CONTACTS AND LOCATIONS:
Overall Officials: Max D Pereira, Phd, Principal Investigator — Federal University of São Paulo; Gabriela PR Prado, MS, Study Chair — Federal University of São Paulo; Fabianne MG Furtado, PhD, Study Chair — Federal University of São Paulo; João PR Biló, MD, Study Chair — Federal University of São Paulo; Lydia M Ferreira, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Prado GP, Pereira MD, Bilo JP, Furtado F, Ferreira LM. Stability of surgically assisted rapid palatal expansion: a randomized trial. J Dent Res. 2013 Jul;92(7 Suppl):49S-54S. doi: 10.1177/0022034513486899. Epub 2013 May 20. PMID 23690355